CLINICAL TRIAL: NCT00259571
Title: Prospektive, Randomisierte, Doppelblinde, Mesalazin-kontrollierte ("Double-dummy Verfahren) Multizenter-Studie Zur Beurteilung Der Annahme Der äquivalenten Wirkung Von Intestinal Retardiert Freigesetztem Phosphatidylcholin gegenüber Mesalazin (Non-inferiority Study) in Der Remissionserhaltung Der Colitis Ulcerosa.
Brief Title: Retarded Phosphatidylcholine Versus Mesalazin in Remission of Ulcerative Colitis.
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Missing financial sponsorship
Sponsor: Heidelberg University (Other)
Collaborators: Dietmar Hopp Stiftung (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PC4; EC - L389/2003; BFARM - 402 2918
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2005-11

CONDITIONS: Ulcerative Colitis
Keywords: remission; mesalazin; non-inferiority study; relapse
MeSH Terms: conditions — Colitis, Ulcerative; Recurrence

INTERVENTIONS:
Drug: retarded release phosphatidylcholine — 2g daily, given orally QTD

SUMMARY:
The purpose of this study is to evaluate if retarded phosphatidylcholine is as effective as mesalazin in preventing an acute episode in ulcerative colitis.

The hypothesis is, that ulcerative colitis is cuased by a defect in the barrier function of the colonic mucus. The background of the study is the finding that the phosphatidylcholine content of the colonic mucus is reduced in patients with ulcerative colitis, in both healthy and inflamed parts of the colon.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ulcerative colitis in remission (CAI 3 or less)
* signed letter of content
* no steroids or immunosupressants in the last 6 weeks
* at least 5 relapses in the last 3 years
* last relapse was 8 months ago or less
* complete colonoscopy at entry

Exclusion Criteria:

* pregnancy or breast feeding
* steroids or immunosuppressants
* acute episode of UC
* condition after complete or partial colektomy
* known intolerance to mesalazin
* severe medical disease other than colitis

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2010-03

PRIMARY OUTCOMES:
rate of relapses
relapse is defined as an increase of the clinical Rachmilewitz index to 5 or more, but at least 3 points over a period of 14 days

SECONDARY OUTCOMES:
time to the first relapse
amount of relapses per year
endoscopic index
histolgical score
life quality
side effects

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Stremmel, Professor, Principal Investigator — Heidelberg University
Locations (1):
- Medical Hospital - University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Stremmel W, Merle U, Zahn A, Autschbach F, Hinz U, Ehehalt R. Retarded release phosphatidylcholine benefits patients with chronic active ulcerative colitis. Gut. 2005 Jul;54(7):966-71. doi: 10.1136/gut.2004.052316. PMID 15951544